CLINICAL TRIAL: NCT03933462
Title: A Study for the Assessment of the Benefits of a Novel Mesh Nebulizer in the Treatment of Patients With Stable COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SRC-RDD-InnospireGo-2018-10458
Record Dates: First submitted 2019-04-12; First posted 2019-05-01 (Actual); Results first posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- InnoSpire Go (Experimental): The InnoSpire Go is a handheld, single patient use, vibrating mesh nebulizer system designed to aerosolize liquid medications for respiratory disease. The device operates continuously once initiated and automatically switches off once the medication has been delivered. The device may be used in pediatric and adult populations, as permitted by the prescribed medication, and is suitable for use in home environments or hospital/clinic settings.
  Interventions: Device: InnoSpire Go
- Jet Nebulizer (Active Comparator): Jet Nebulizers are the standard delivery system for aerosolized medications. A nebulizer breaks up medical solutions into small droplets suspended in air (aerosol) so that they may be delivered to the patient's airways for respiratory therapy.
  Interventions: Device: Jet Nebulizer

INTERVENTIONS:
Device: InnoSpire Go — Participants will use for 30 days.
  Arms: InnoSpire Go
Device: Jet Nebulizer — Participants will use for 30 days.
  Arms: Jet Nebulizer

SUMMARY:
Jet nebulizers have been the standard delivery system for aerosolized medications commonly prescribed to Chronic Obstructive Pulmonary Disease (COPD) patients; however, these devices are inefficient and require an external pressurized gas source to operate. Vibrating mesh nebulizers have a significantly higher efficiency of delivering drugs to the lung compared to conventional jet or ultrasonic nebulizers because of the high fine particle fraction created by the rapid vibration. This post-market study will investigate the potential benefits of a vibrating mesh nebulizer compared a standard jet nebulizer. The study will include stable, ambulatory COPD patients who are currently using a jet nebulizer system. Participants will be asked to use each device for a period of 30 days. Patient preference and changes to quality of life will be evaluated.

DETAILED DESCRIPTION:
Participants will be contacted by designated study site staff. Participants may be pre-screened through medical records over the phone to assess potential eligibility. A screening script will include a general review of key inclusion and exclusion criteria. Participants that are interested will be scheduled for a screening visit at the clinical office.

Visit 1 - Screening/Baseline:

Once the participant arrives, the study will be explained in full detail. If the participant agrees, he/she will be consented into the study and the participant will be given a copy of the informed consent. After the consent is signed, the following procedures will be performed:

Demographics

Medical History

Concomitant Medication

mMRC

Chronic Respiratory Disease Questionnaire (CRQ) Self-Reported (SR)

Pulmonary Function Tests

Vital Signs prior to 6 Minute Walk (6MW)

6-Minute Walk Test (6MWT)

Modified Borg Assessment

Inclusion/Exclusion Criteria Review

Device Photograph

Randomization Participants will be randomly assigned to either their current jet nebulizer or the InnoSpire Go device for the first 30 days of treatment.

Training Session Participants randomized to InnoSpire Go in the first treatment arm will be trained on the use and cleaning of the device before being sent home.

Visit 2 - Interim Visit:

Participants will be asked to return to the research center 15 days ± 3 days after Visit 1.

Side Effect and Adverse Event Assessment Participants will be asked about any side effects or adverse events (AEs) since the last visit.

Concomitant Medications

CRQ-SR (Follow-Up)

Nebulizer Satisfaction Assessment Participant satisfaction with the device used in the first treatment arm will be assessed.

Visit 3 - Cross-over:

Participants will be asked to return to the research center within 30 days ± 3 days after Visit 1. They will be instructed to bring the first assigned study device and their prescribed albuterol or combination albuterol/ipratropium medication for the demonstration.

CRQ-SR (Follow-Up)

Concomitant Medications

Device Use Demonstration

Nebulizer Weight The nebulizer cup/reservoir alone will be weighed with the medication before device use and after device use to capture residual medication. This process will take place during video recording.

Peak inspiratory flow (PIF)

Vital Signs prior to 6MW

. Modified Borg Assessment

6-Minute Walk Test

Nebulizer Satisfaction Assessment Participant satisfaction with the device used in the first treatment arm will be assessed.

Training Session Participants randomized to InnoSpire Go in the second treatment arm will be trained on the use and cleaning of the device before being sent home.

Visit 4 - Interim Visit:

Participants will be asked to return to the research center 15 days ± 3 days after Visit 3. Participants will complete procedures outlined in Visit 2.

Visit 5 -Final Visit:

Participants will return to the clinical facility 30 days (± 3 days) after Visit 3 completion. They will be instructed to bring the second assigned study device and their prescribed albuterol or combination albuterol/ipratropium medication for the demonstration. Participants will complete the procedures outlined in Visit 3. Participants will need to return all study equipment at this visit.

Participants will be discharged from the study following completion of study procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 40 years of age.
2. Diagnosis of COPD.
3. Currently using only a mouthpiece with their nebulizer system.
4. Forced Expiratory Volume at 1 second (FEV1) ≥ 30% predicted (pre or post bronchodilator).
5. Modified Medical Research Council (mMRC) Dyspnea scale grade ≥ 1.
6. Use of a jet nebulizer for the administration of albuterol or combination albuterol/ipratropium for the past 6 months
7. Willing to use the same compressor/nebulizer system throughout the study
8. Willing to refrain from using the jet nebulizer system when using InnoSpire Go
9. Prescribed nebulizer combination albuterol/ipratropium (single or multiple vials) with self-report of at least daily use or prescribed nebulizer albuterol with self-report of at least twice daily use.
10. Willing to permit audio and video recording during the visit.
11. Willing and able to follow instructions and complete all activities required by the trial, including phone calls.
12. Able to read and understand English.

Exclusion Criteria:

1. Unable to complete 6MWT or, if patient is not currently prescribed oxygen, persistent oxygen desaturation ≤ 88% on the 6MWT.
2. Exacerbation of COPD requiring hospitalization in the last 3 months (defined as hospital admission, urgent care visit, or emergency room visit).
3. Prescribed non-selective beta blockers.
4. Prescribed additional ipratropium bromide via nebulizer or inhaler or any other nebulized treatments via the subject's jet nebulizer.
5. Patients currently in assisted living or nursing home.
6. Diagnosis of asthma, parenchymal lung disease other than COPD, bronchiectasis, tuberculosis, cor pulmonale, clinically significant obstructive urinary disease, narrow-angle glaucoma, unstable angina, depression, anxiety, or other serious medical condition that, in the opinion of the investigator, would interfere with the patient's participation in the trial.
7. History of thoracotomy.
8. Myocardial infarction within the last 6 months.
9. Participation in any other therapeutic clinical trial in the previous 4 weeks

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2019-10-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Jefferson Associates in Internal Medicine,LTD, Clairton, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nickerson C, Hollen DV, Garbin S, Doty K, Jasko J, Cain C. Pilot Study to Investigate the Benefits of the InnoSpire Go Mesh Nebulizer Compared to Jet Nebulizers in the Treatment of Stable COPD. J Aerosol Med Pulm Drug Deliv. 2022 Aug;35(4):186-195. doi: 10.1089/jamp.2021.0054. Epub 2022 Feb 23. PMID 35196114

RESULTS

PARTICIPANT FLOW:
Groups:
- InnoSpire Go, Then Current Jet Nebulizer: Participants first assigned to use the InnoSpire Go for nebulizer treatments for 30 days. Then they then were assigned to use their current jet nebulizer for nebulizer treatments for 30 days
- Current Jet Nebulizer, Then Innospire Go: Participants first assigned to use their current jet nebulizer for nebulizer treatments for 30 days. Then they then were assigned to use Innospire Go for nebulizer treatments for 30 days.
Period: Overall Study
Arm/Group | InnoSpire Go, Then Current Jet Nebulizer | Current Jet Nebulizer, Then Innospire Go
Started | 10 | 10
Crossover | 8 | 10
Completed | 8 | 10
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants that signed a consent form.
Arm/Group | All Participants
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21
Body Mass Index(BMI) [Mean (Standard Deviation); unit: kilograms/m^2] | 27.8 (6.8)

OUTCOME MEASURES:

1. Primary Outcome: Device Preference Among the Number of Participants.
Description: Device preference after 60 days of device use as determined by the nebulizer satisfaction questionnaire in stable ambulatory Chronic Obstructive Pulmonary Disease (COPD) patients.
  The nebulizer satisfaction questionnaire is an 11 question survey developed to determine device satisfaction. 10 questions are answered on a scale of 0 to 10 with 0 being the worst and 10 being the best. The last question in the survey is in regards to device preference and is only asked at the end of the study.
Time Frame: 60 days
Population: One participant removed from the data set because they were on the incorrect standard of care device.
Measure: Count of Participants; unit: Participants
Arm/Group | InnoSpire Go | Jet Nebulizer
Number analyzed (Participants) | 17 | 17
Participants | 17 | 0
Statistical Analysis 1: Comparison: InnoSpire Go vs Jet Nebulizer; Test type: Superiority — Categorical preference endpoints that answered at the final visit (e.g., "Which device do you prefer?") were analyzed with a One-sample Binomial Test that compared the observed proportion to a 50/50 split; p < 0.001, One Sample Binomial

2. Secondary Outcome: Change in Quality of Life From Baseline on the CRQ-SR
Description: Change in quality of life scores (mean difference) after 30 days of each device use compared to baseline as determined by the Chronic Respiratory disease Questionnaire - Self-Report (CRQ-SR). The scores for each question in each dimension are simply added together. Using a seven-point scale for the responses, the minimum and maximum scores for each dimension are as follows: Minimum score Maximum score (Worst function is 1) (Best function is 7)
Time Frame: baseline and 30 days for each intervention
Population: One participant removed from the data set because they were on the incorrect standard of care device.
Measure: Mean (Standard Deviation); unit: mean difference of units on a scale
Arm/Group | InnoSpire Go | Jet Nebulizer
Number analyzed (Participants) | 17 | 17
mean difference of units on a scale
  Dyspnea | 1.2 (2.1) | 0.8 (2.1)
  Fatigue | 0.7 (1.9) | 0.2 (1.9)
  Emotional Function | 0.6 (1.5) | 0.1 (1.5)
  Mastery | 0.8 (1.6) | 0.1 (1.6)

3. Other Pre Specified Outcome: Difference in Total Distance Walked as Measured by a 6-Minute Walk Test
Description: Difference in total distance walked as measured by a 6-Minute Walk Test (6MWT) between participants jet nebulizer and InnoSpire Go
Time Frame: 30 days, 30 days
Population: One participant removed from the data set because they were on the incorrect standard of care device.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | InnoSpire Go | Jet Nebulizer
Number analyzed (Participants) | 17 | 17
meters | 278.7 (111.0) | 275.7 (125.6)

4. Other Pre Specified Outcome: Change in Modified Borg Score
Description: The change in the modified Borg score following 6MWT, where the visit's post-nebulizer Borg score will be used as the baseline for this endpoint. The change in the modified Borg score following nebulizer use, where the visit's pre-nebulizer Borg score will be used as the baseline for this endpoint. Difference in modified Borg score from pre-nebulizer to post-6MWT for each device. This is a scale that asks you to rate the difficulty of your breathing. It starts at number 0 where your breathing is causing you no difficulty at all and progresses through to number 10 where your breathing difficulty is maximal.
Time Frame: 30 days, 30 days
Population: One participant removed from the data set because they were on the incorrect standard of care device.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | InnoSpire Go | Jet Nebulizer
Number analyzed (Participants) | 17 | 17
score on a scale
  Borg: 15 Min After Neb/Borg: Before Neb Use | -1.32 (0.86) | -1.09 (0.48)
  Borg: After 6MWT/Borg: 15 Min After Neb Use | 6.38 (1.57) | 7.09 (1.38)
  Borg: After 6MWT/Borg: Before Neb Use | 5.06 (2.00) | 6.00 (1.25)

5. Other Pre Specified Outcome: Participant Satisfaction Based on Specific Elements of the Device's Operation and Handling
Description: Difference in device confidence, perceived effect, difficulty of device assembly/disassembly, difficulty of cleaning and regular care, overall ease of handling or usability, overall burden, medication delivery confidence, overall satisfaction, likelihood of recommending, perception of with lifestyle and average ease of use score after each 30 days of device use. This assessment is a 10 question survey were respondents answer questions on a scale 0 to 10 with 0 being the worse and 10 being the best. Each question has a score of 0 to 10.
Time Frame: 30 days, 30 days
Population: One participant removed from the data set because they were on the incorrect standard of care device.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | InnoSpire Go | Jet Nebulizer
Number analyzed (Participants) | 17 | 17
score on a scale
  Confidence with use | 9.6 (0.8) | 7.9 (2.8)
  Effect on shortness of breath | 8.8 (1.7) | 6.9 (1.9)
  Difficulty of assembly/disassembly | 9.9 (0.5) | 7.1 (2.9)
  Difficulty of Cleaning | 9.6 (0.9) | 7.2 (2.9)
  Overall usablity | 9.4 (2.2) | 6.5 (2.9)
  Overall Burden | 9.6 (1.1) | 5.8 (3.1)
  Confidence in medication delivery | 9.8 (1.0) | 6.4 (3.1)
  Overall Satisfaction | 9.2 (2.4) | 5.9 (2.8)
  Likelihood recomendation | 9.9 (0.5) | 5.1 (3.2)
  Fit with Lifestyle | 9.8 (1.0) | 4.4 (2.7)

6. Other Pre Specified Outcome: Difference in Participant Use Time
Description: Time spent using the device will be compared between each device. The following times will be analyzed:
  Time in mouth (treatment time = first insert of mouthpiece to last removal of mouthpiece)
Time Frame: 30 days, 30 days
Population: One participant did not have video data for InnospireGo and was excluded for the analysis.,
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | InnoSpire Go | Jet Nebulizer
Number analyzed (Participants) | 16 | 16
minutes | 5.0 (0.7) | 9.1 (5.8)

7. Other Pre Specified Outcome: Amount of Fluid Nebulized
Description: Amount of fluid nebulized (pre- and post-weight of nebulizer) between each device
Time Frame: 30 days, 30 days
Population: One participant removed from the data set because they were on the incorrect standard of care device.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | InnoSpire Go | Jet Nebulizer
Number analyzed (Participants) | 17 | 17
grams | -2.4 (0.3) | -2.1 (0.7)

8. Other Pre Specified Outcome: Difference in Participant Time to Fill
Description: Time spent using the device will be compared between each device. The following time will be analyzed:
  Time to fill (open disposable nebulizer, dispense ampule, close or reassemble)
Time Frame: 30 days, 30 days
Population: Difficult to discern due to poor video quality.
Arm/Group | InnoSpire Go | Jet Nebulizer
Number analyzed (Participants) | 0 | 0

9. Other Pre Specified Outcome: Difference in Participant Time to Sputter
Description: Time spent using the device will be compared between each device. The following time will be analyzed:
  Time to sputter.
Time Frame: 30 days, 30 days
Population: Difficult to standardized as it is difficult to hear and observed aerosol mist with the different jet nebulizers
Arm/Group | InnoSpire Go | Jet Nebulizer
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 60 days
Groups:
- InnoSpire Go: Participants first assigned to use the InnoSpire Go for nebulizer treatments for 30 days.
- Jet Nebulizer: Participants first assigned to use their current jet nebulizer for nebulizer treatments for 30 days.
Arm/Group | InnoSpire Go | Jet Nebulizer
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 2/21 | 0/21
Other Adverse Events (participants affected / at risk) | 1/21 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | InnoSpire Go (N=21) | Jet Nebulizer (N=21)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | InnoSpire Go (N=21) | Jet Nebulizer (N=21)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-07): https://cdn.clinicaltrials.gov/large-docs/62/NCT03933462/Prot_SAP_000.pdf